CLINICAL TRIAL: NCT04656938
Title: Promoting Health LongevIty Through Mitigation and Prevention of Frailty in Community-dwelling Elderly (Pro-LIFE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/2353
Record Dates: First submitted 2020-11-19; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Frailty; Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: This is a pre-post study design with a single group and no control arm. The study aims to screen 700 participants, of which, 220 pre-frail seniors to be recruited into the intervention programme.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pre-frail intervention — Pre-frail partiipants will undergo 4 month intervention consisted of group-based physical exercise and nutritional classes.

SUMMARY:
The current healthcare response to frailty has been mainly reactive to acute health crises of the elderly. With its insidious onset and progression, frailty is often not apparent unless actively sought. Well-validated models of frailty already exist and, instead of trying to create new frailty criteria or insisting on a universal approach to measuring frailty, it is needed to move on to higher levels of care systems supporting their practical implementation, mapping the chosen frailty instrument to its specific role. This pragmatic study will equip older persons with awareness of their frailty status through community-based screening, allowing for timely stage-specific care to avoid deleterious outcomes. While older persons meeting frailty criteria will be referred for comprehensive geriatric assessment, pre-frail older persons will be targeted for multi-factorial exercise and nutritional intervention in the community to reverse the frailty trajectory. An over-arching aim will be to create a sustainable triaging system and early intervention programme that can be administered by trained members of the community. This will allow older persons to receive regular re-assessments in the community such that any transitions to a higher state of frailty may be captured and promptly addressed.

DETAILED DESCRIPTION:
This is a non-controlled prospective cohort study, recruiting community-dwelling older persons aged >55 years, from various senior activity centres, day care and community centres in the North-East region of Singapore. A mobile community-based platform for frailty and physical fitness assessment will be anchored at the void decks of public housing blocks, senior activity centres (SACs), senior care centres (SCCs) or community clubs for accessibility. The platform will be maintained at each site for 2-3 consecutive weeks, and is managed by members of the multidisciplinary team, with the same site being re-visited at yearly intervals to allow follow-up. Each participant undergoes a multi-domain geriatric screen and physical fitness assessment, and will be triaged by physical frailty status for stage-specific care.

Written informed consent will be obtained from all participants, and ethics approval has been obtained from the Institutional Review Board of Singhealth.

Measures Multi-domain geriatric screen The multi-domain geriatric screen includes assessment of (i) socio-demographic characteristics (including social support network, socio-economic status, education and employment); (ii) mood as assessed using the 15-item Geriatric Depression Scale; (iii) cognitive performance using the locally validated modified Chinese version of Mini Mental State Examination (CMMSE); (iv) nutrition using the Mini Nutrition Assessment-Short Form (MNA-SF) and Subjective Global Assessment (SGA); (iv) physical activity level based on a structured questionnaire to assess the time spent on physical activities over the last 7 days; (v) functional performance using Barthel's Index for activities of daily living (ADLs) and Lawton and Brody's instrumental ADLs, as well as Life Space Questionnaire (LSQ) for functional mobility; (vi) quality of life on EuroQol 5 dimensions (EQ-5D-5L) questionnaire and a visual analogue scale; (vii) sarcopenia using SARC-F questionnaire enquiring ability to carry a heavy load, walking, rising from a chair, climbing stairs and falls, has been validated as a suitable tool for community screening for sarcopenia.

Frailty Assessment Frailty screening will be based on the 5-item FRAIL scale, which assesses for self-reported fatigue, resistance, ambulation, illnesses and loss of weight, to categorize participants as frail (score 3-5), pre-frail (1-2) or robust (0).

Physical frailty will be objectively assessed using modified Fried's criteria, with frailty defined by the presence of at least 3 and pre-frailty as 1-2 of 5 components - exhaustion, slow gait speed, weak grip strength, low body mass index (BMI<18.5kg/m2) and low physical activity.

Grip strength will be measured using a JAMAR hand dynamometer, with 2 trials for each hand, and the maximum value will be used for analysis. Gait speed will be based on time taken to walk 10m at usual pace. Weakness (<18kg for women and <26 kg for men) and slowness (<0.8m/s) will be defined using reference values from the Asian Working Group for Sarcopenia

Physical Fitness Tests The physical fitness test battery was modified from the Senior Fitness Test. Participants who report feeling unwell on pre-assessment screening will be exempt from fitness tests.

Lower body strength and power will be measured using the chair stand test, in which the participant will be instructed to rise as fast as possible from seated to a full standing position, while keeping the arms folded across the chest. Time taken to complete 5 chair stands as well as the number of full chair stands performed in 30 seconds will be recorded.

In addition to grip strength, upper limb dexterity will be assessed using the box-and-block test, in which participants pick up blocks and place them in the box on the other side across a barrier as quickly as possible. The number of blocks transferred in 1 minute will be recorded. 2 trials will be performed, one for each arm, and the better performance will be used for analysis.

Dual-task gait performance will be assessed by asking the participant to walk 10-metres while performing serial 2-step forward calculation and animal naming without specific instruction on task prioritization. Gait speed and number of correct calculations on the dual-task protocol will be recorded.

Upper and lower body flexibility will be assessed using the back-scratch and chair sit-and-reach tests respectively, with 2 trials for each test, and the better performance will be used for analysis. The back-scratch test is performed with the participant placing one hand behind the shoulder and the other hand up the middle of the back, fingers extended. The distance (cm) the middle fingers are short of touching (-) or overlapping (+) will be recorded. In the chair sit-and-reach test, participant sits on the edge of a chair with one leg extended in front while reaching forward with the hands toward the toes. The distance (cm) from the extended third finger to tip of toe (+ for beyond, and - for behind the toe) will be recorded.

Dynamic balance (agility) will be assessed on the Timed Up-and-Go Test, which requires the participant to stand from a seated position, walk as quickly as possible around a cone 3m ahead of the chair, and return to a fully seated position. The balance subtests of the Short Physical Performance Battery (SPPB) was also adopted, including side-by-side, semi-tandem and tandem standing.

Cardiorespiratory endurance will be evaluated using the 6-minute walk test (6MWT), along a walkway of at least 20m and with constant encouragement throughout the test. The total distance walked in 6 minutes will be recorded, and rest is permitted anytime during the test.

Each participant will be scored on the SPPB for a composite measure of physical performance, applying established cut-offs on the individual tests of gait speed, balance and chair stand.

Body Composition Participants will under Bioimpedance Analysis (BIA) (MC-780M, TANITA, Tokyo, Japan) for measurement of muscle mass.

Intervention for pre-frail older adults Pre-frail will be operationalized as the presence of 1-2 positive responses on FRAIL, or FRAIL score of 0 but with objective weak grip strength and/or slow gait speed. The latter takes into consideration the potential for under-reporting of symptoms on the FRAIL questionnaire.

Participants meeting operational criteria for pre-frailty will be enrolled in a group-based physical exercise and nutritional intervention programme, delivered over 4 months. The intervention will commence 3 months from the baseline screening.

Group-based, as opposed to traditional individual physiotherapy sessions, has been shown to boost older persons' motivation for participation and potentially addresses the social contribution to frailty.

Participants will undergo weekly 1-hr exercise sessions designed to challenge all major muscle groups with specific emphasis on strength training, in addition to gait, balance and endurance exercises, to target the major frailty elements of weakness and gait deficit, with demonstrated effectiveness for falls prevention in older adults. Upper limb strengthening exercises will be conducted through the use of therabands or free weights (e.g. bottled water) for resistance. The exercises will be made progressively more difficult over time (e.g. increasing the number of repetitions) according to group's progress, yet also catering for individual variability, under supervision of the physiotherapist. Endurance exercise will consist of outdoor walking. Targeting to each older adult's individual intensity level with progression as they improve ensures that the exercises remain physically challenging to provide sufficient stimulus. An individually prescribed structured home exercise programme with pictorials and explanations at the end of each session will be provided so that participants can continue with the exercises between sessions to achieve an optimal frequency of exercising at least three times a week, with a checklist to record adherence.

Nutritional intervention (6 group-based session) will be delivered with the aim of facilitating healthy eating habits to achieve adequate protein, energy, Vitamin D and fluid intake through regular foods and beverages without the need for nutritional supplements. Educating older adults to evaluate and adapt their nutritional intake, taking into consideration their dietary habits, can be expected to improve sustainability of effect and adherence. A group grocery-shopping trip will be conducted to provide guidance on choosing quality food within budget.

All participants will be followed up at 6-, 12- and 24-month. Participants enrolled in the intervention programme will have their physical performance measures at 3-month (immediate pre-intervention). Subsequent follow-up visits will be at the end of the 4-month intervention, 6- and 12-month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* any community-dwelling adult aged 55 and above
* able to ambulate independently (use of walking aids permitted)

Exclusion Criteria:

* For the pre-frail intervention programme, older adults with significant cognitive impairment, as defined using age- and education-adjusted local norms on the modified Chinese version of the Mini-Mental State Examination (CMMSE) will be excluded

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Frailty Prevalence in Community-dwelling older adults | Baseline
  Prevalence of pre-frailty and frailty in community-dwelling older adults aged >55 years who attend frailty screening. Frailty will be measured using the 5-item FRAIL questionnaire, which assesses for self-reported fatigue, resistance, ambulation, illnesses and loss of weight. 1 point is assigned for each positive response, and participants are categorized as frail (score 3-5), pre-frail (1-2) or robust (0). Agreement of the FRAIL scale with established frailty measures - Fried Phenotype and Frailty Index (35-item) will be examined.
Proportion of pre-frail participant reverting to robustness following a 4-month multi-factorial physical exercise and nutrition intervention programme | End of intervention (7-month)
  For intervention eligibility, pre-frailty will be operationalized as: (i) FRAIL score 1-2, or (ii) FRAIL score 0 but with weak grip strength or slow gait speed based on Asian Working Group for Sarcopenia cut-offs. The proportion of pre-frail participants who revert to being robust at the end of the 4-month intervention programme will be measured.
Change in physical performance measures among pre-frail older adults following a 4-month exercise and nutrition intervention programme | End of intervention (7-month)
  Physical performance measures include grip strength, gait speed (time taken to 10-m walk at usual pace), lower limb strength (time taken to complete 5 chair stands and number of chair stands completed in 30-seconds), upper and lower limb flexibility (back-scratch test and modified sit-and-reach test), upper limb dexterity (box-and-block test), tandem and dynamic balance (Timed-Up-and-Go test), and cardiorespiratory endurance (6-minute walk test). Cut-off values for tests of gait speed, balance and chair-stand will be applied to derive a score on the Short Physical Performance Battery as a composite measure of physical performance.

SECONDARY OUTCOMES:
Performance in physical fitness tests at 3 month (immediate pre-intervention) | 3-month
  Physical performance measures include grip strength, gait speed (time taken to 10-m walk at usual pace), lower limb strength (time taken to complete 5 chair stands and number of chair stands completed in 30-seconds), upper and lower limb flexibility (back-scratch test and modified sit-and-reach test), upper limb dexterity (box-and-block test), tandem and dynamic balance (Timed-Up-and-Go test), and cardiorespiratory endurance (6-minute walk test). Cut-off values for tests of gait speed, balance and chair-stand will be applied to derive a score on the Short Physical Performance Battery as a composite measure of physical performance.
Performance in physical fitness tests at 7-month (immediate post-intervention) | 7-month
  Physical performance measures include grip strength, gait speed (time taken to 10-m walk at usual pace), lower limb strength (time taken to complete 5 chair stands and number of chair stands completed in 30-seconds), upper and lower limb flexibility (back-scratch test and modified sit-and-reach test), upper limb dexterity (box-and-block test), tandem and dynamic balance (Timed-Up-and-Go test), and cardiorespiratory endurance (6-minute walk test). Cut-off values for tests of gait speed, balance and chair-stand will be applied to derive a score on the Short Physical Performance Battery as a composite measure of physical performance.
Performance in physical fitness tests at 13-month (6 months post-intervention) | 13-month
  Physical performance measures include grip strength, gait speed (time taken to 10-m walk at usual pace), lower limb strength (time taken to complete 5 chair stands and number of chair stands completed in 30-seconds), upper and lower limb flexibility (back-scratch test and modified sit-and-reach test), upper limb dexterity (box-and-block test), tandem and dynamic balance (Timed-Up-and-Go test), and cardiorespiratory endurance (6-minute walk test). Cut-off values for tests of gait speed, balance and chair-stand will be applied to derive a score on the Short Physical Performance Battery as a composite measure of physical performance.
Performance in physical fitness tests at 19-month (12 months post-intervention) | 19-month
  Physical performance measures include grip strength, gait speed (time taken to 10-m walk at usual pace), lower limb strength (time taken to complete 5 chair stands and number of chair stands completed in 30-seconds), upper and lower limb flexibility (back-scratch test and modified sit-and-reach test), upper limb dexterity (box-and-block test), tandem and dynamic balance (Timed-Up-and-Go test), and cardiorespiratory endurance (6-minute walk test). Cut-off values for tests of gait speed, balance and chair-stand will be applied to derive a score on the Short Physical Performance Battery as a composite measure of physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tay, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No